CLINICAL TRIAL: NCT01029236
Title: The Effect of Metabolism-Boosting Beverages on 24 Hr Energy Expenditure
Brief Title: Evaluation of Metabolism-Boosting Beverages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medifast, Inc. (Industry)
Responsible Party: Lisa M. Davis, PhD, PA-C/ Vice President of Research and Development, Medifast Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MED010; 20070530 (Other: Western Institutional Review Board)
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Energy Expenditure; Appetite
Keywords: obesity; metabolism; weight loss; energy expenditure; thermogenesis; Metabolism-Boosting Beverages effect on REE; Metabolism-Boosting Beverages effect on appetite
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Medifast Metabolism-boosting Beverages — Medifast metabolism-boosting beverages containing 90 mg EGCG and 100 mg caffeine.

SUMMARY:
The purpose of this study is to assess the effect of Metabolism-boosting Beverages (MBB) containing green tea extract with a standardized amount of epigallocatechin gallate (EGCG) and caffeine.

DETAILED DESCRIPTION:
The study will assess the effect of MBB's on 24 hour energy expenditure by performing indirect calorimetry, and on appetite using visual analogue scales (VAS). The planned sample size is 54 healthy male and female adults, both lean and overweight. We plan to test 6 metabolism-boosting beverages in the following order: 1) Raspberry Tea 2) Banana Shake 3) Chai Latte 4) Strawberry Shake 5) Cappuccino 6) Hot Cocoa. In the order that they are screened, each subject will be assigned to receive 1 of 6 Metabolism-boosting beverages. Each MBB will contain 90 mg EGCG and 100 mg caffeine.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females (age between 18 and 65)
* BMI ≥18.5 - ≤ 40.0 kg/m2
* Non-smokers
* No known food allergies to wheat, gluten, soy or nuts
* ≤ 14 alcoholic beverages per week
* No sensitivity to caffeine or green tea
* No alcohol or caffeine on days when metabolism is tested
* Willing and able to give informed consent
* Not currently using appetite-affecting medications (e.g SSRIs, steroids, Ritalin)
* Not pregnant or lactating

Exclusion Criteria:

* Actively dieting
* Chronic uncontrolled health problems (not including obesity or controlled: type-2 diabetes, hyperlipidemia, hypertension)
* History of arrhythmia, or taking anti-arrhythmic medications (e.g. propafenone)
* Schizophrenia, history of bipolar disorder, current Major Depressive Disorder
* Dependence on alcohol or sedative-hypnotic drugs (e.g. benzodiazepines)
* Cognitive impairment severe enough to preclude informed consent
* Taking weight loss or appetite-suppressant medications
* Taking appetite affecting medications (e.g. SSRIs, steroids, Ritalin)
* Food allergies to wheat, gluten, soy, or nuts
* Sensitivity to caffeine or green tea

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To assess the effect of MBBs on REE by performing indirect calorimetry | 30, 60, 90, and 120 minutes

SECONDARY OUTCOMES:
To assess the effect of MBBs on appetite via visual analogue scales | 30, 60, 90, and 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Davis, PhD, PA-C, Principal Investigator — Medifast, Inc.; Christopher D Coleman, MS,RD,LDN, Study Director — Medifast, Inc.
Locations (1):
- Medifast Inc., Owings Mills, Maryland, United States

REFERENCES:
- [Background] Berube-Parent S, Pelletier C, Dore J, Tremblay A. Effects of encapsulated green tea and Guarana extracts containing a mixture of epigallocatechin-3-gallate and caffeine on 24 h energy expenditure and fat oxidation in men. Br J Nutr. 2005 Sep;94(3):432-6. doi: 10.1079/bjn20051502. PMID 16176615
- [Background] Acheson KJ, Schutz Y, Bessard T, Anantharaman K, Flatt JP, Jequier E. Glycogen storage capacity and de novo lipogenesis during massive carbohydrate overfeeding in man. Am J Clin Nutr. 1988 Aug;48(2):240-7. doi: 10.1093/ajcn/48.2.240. PMID 3165600
- [Background] Golay A, Schutz Y, Meyer HU, Thiebaud D, Curchod B, Maeder E, Felber JP, Jequier E. Glucose-induced thermogenesis in nondiabetic and diabetic obese subjects. Diabetes. 1982 Nov;31(11):1023-8. doi: 10.2337/diacare.31.11.1023. No abstract available. PMID 6757011
- [Background] Segal KR, Albu J, Chun A, Edano A, Legaspi B, Pi-Sunyer FX. Independent effects of obesity and insulin resistance on postprandial thermogenesis in men. J Clin Invest. 1992 Mar;89(3):824-33. doi: 10.1172/JCI115661. PMID 1541675
- [Background] den Besten C, Vansant G, Weststrate JA, Deurenberg P. Resting metabolic rate and diet-induced thermogenesis in abdominal and gluteal-femoral obese women before and after weight reduction. Am J Clin Nutr. 1988 May;47(5):840-7. doi: 10.1093/ajcn/47.5.840. PMID 3364400
- [Background] Abbott RD, Ross GW, White LR, Nelson JS, Masaki KH, Tanner CM, Curb JD, Blanchette PL, Popper JS, Petrovitch H. Midlife adiposity and the future risk of Parkinson's disease. Neurology. 2002 Oct 8;59(7):1051-7. doi: 10.1212/wnl.59.7.1051. PMID 12370461
- [Background] Allison DB, Gadbury G, Schwartz LG, Murugesan R, Kraker JL, Heshka S, Fontaine KR, Heymsfield SB. A novel soy-based meal replacement formula for weight loss among obese individuals: a randomized controlled clinical trial. Eur J Clin Nutr. 2003 Apr;57(4):514-22. doi: 10.1038/sj.ejcn.1601587. PMID 12700612
- [Background] Borchardt RT, Huber JA. Catechol O-methyltransferase. 5. Structure-activity relationships for inhibition by flavonoids. J Med Chem. 1975 Jan;18(1):120-2. doi: 10.1021/jm00235a030. No abstract available. PMID 1109569
- [Background] Curatolo PW, Robertson D. The health consequences of caffeine. Ann Intern Med. 1983 May;98(5 Pt 1):641-53. doi: 10.7326/0003-4819-98-5-641. PMID 6342491
- [Background] Diepvens K, Westerterp KR, Westerterp-Plantenga MS. Obesity and thermogenesis related to the consumption of caffeine, ephedrine, capsaicin, and green tea. Am J Physiol Regul Integr Comp Physiol. 2007 Jan;292(1):R77-85. doi: 10.1152/ajpregu.00832.2005. Epub 2006 Jul 13. PMID 16840650
- [Background] Dulloo AG. Ephedrine, xanthines and prostaglandin-inhibitors: actions and interactions in the stimulation of thermogenesis. Int J Obes Relat Metab Disord. 1993 Feb;17 Suppl 1:S35-40. PMID 8384178
- [Background] Dulloo AG, Duret C, Rohrer D, Girardier L, Mensi N, Fathi M, Chantre P, Vandermander J. Efficacy of a green tea extract rich in catechin polyphenols and caffeine in increasing 24-h energy expenditure and fat oxidation in humans. Am J Clin Nutr. 1999 Dec;70(6):1040-5. doi: 10.1093/ajcn/70.6.1040. PMID 10584049
- [Background] Festi D, Colecchia A, Sacco T, Bondi M, Roda E, Marchesini G. Hepatic steatosis in obese patients: clinical aspects and prognostic significance. Obes Rev. 2004 Feb;5(1):27-42. doi: 10.1111/j.1467-789x.2004.00126.x. PMID 14969505
- [Background] Gale SM, Castracane VD, Mantzoros CS. Energy homeostasis, obesity and eating disorders: recent advances in endocrinology. J Nutr. 2004 Feb;134(2):295-8. doi: 10.1093/jn/134.2.295. PMID 14747663
- [Background] Gougeon R, Harrigan K, Tremblay JF, Hedrei P, Lamarche M, Morais JA. Increase in the thermic effect of food in women by adrenergic amines extracted from citrus aurantium. Obes Res. 2005 Jul;13(7):1187-94. doi: 10.1038/oby.2005.141. PMID 16076988
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] Heymsfield SB, van Mierlo CA, van der Knaap HC, Heo M, Frier HI. Weight management using a meal replacement strategy: meta and pooling analysis from six studies. Int J Obes Relat Metab Disord. 2003 May;27(5):537-49. doi: 10.1038/sj.ijo.0802258. PMID 12704397
- [Background] Keaney JF Jr, Larson MG, Vasan RS, Wilson PW, Lipinska I, Corey D, Massaro JM, Sutherland P, Vita JA, Benjamin EJ; Framingham Study. Obesity and systemic oxidative stress: clinical correlates of oxidative stress in the Framingham Study. Arterioscler Thromb Vasc Biol. 2003 Mar 1;23(3):434-9. doi: 10.1161/01.ATV.0000058402.34138.11. Epub 2003 Jan 30. PMID 12615693
- [Background] Klaus S, Pultz S, Thone-Reineke C, Wolfram S. Epigallocatechin gallate attenuates diet-induced obesity in mice by decreasing energy absorption and increasing fat oxidation. Int J Obes (Lond). 2005 Jun;29(6):615-23. doi: 10.1038/sj.ijo.0802926. PMID 15738931
- [Background] Pouliot MC, Despres JP, Nadeau A, Moorjani S, Prud'Homme D, Lupien PJ, Tremblay A, Bouchard C. Visceral obesity in men. Associations with glucose tolerance, plasma insulin, and lipoprotein levels. Diabetes. 1992 Jul;41(7):826-34. doi: 10.2337/diab.41.7.826. PMID 1612197
- [Background] Fiorini RN, Donovan JL, Rodwell D, Evans Z, Cheng G, May HD, Milliken CE, Markowitz JS, Campbell C, Haines JK, Schmidt MG, Chavin KD. Short-term administration of (-)-epigallocatechin gallate reduces hepatic steatosis and protects against warm hepatic ischemia/reperfusion injury in steatotic mice. Liver Transpl. 2005 Mar;11(3):298-308. doi: 10.1002/lt.20348. PMID 15719408
- [Background] Rumpler W, Seale J, Clevidence B, Judd J, Wiley E, Yamamoto S, Komatsu T, Sawaki T, Ishikura Y, Hosoda K. Oolong tea increases metabolic rate and fat oxidation in men. J Nutr. 2001 Nov;131(11):2848-52. doi: 10.1093/jn/131.11.2848. PMID 11694607
- [Background] Segal KR, Gutin B, Nyman AM, Pi-Sunyer FX. Thermic effect of food at rest, during exercise, and after exercise in lean and obese men of similar body weight. J Clin Invest. 1985 Sep;76(3):1107-12. doi: 10.1172/JCI112065. PMID 4044828
- [Background] Rudelle S, Ferruzzi MG, Cristiani I, Moulin J, Mace K, Acheson KJ, Tappy L. Effect of a thermogenic beverage on 24-hour energy metabolism in humans. Obesity (Silver Spring). 2007 Feb;15(2):349-55. doi: 10.1038/oby.2007.529. PMID 17299107
- [Background] Thearle M, Aronne LJ. Obesity and pharmacologic therapy. Endocrinol Metab Clin North Am. 2003 Dec;32(4):1005-24. doi: 10.1016/s0889-8529(03)00066-5. PMID 14711072
- [Background] Westerterp-Plantenga MS, Lejeune MP, Kovacs EM. Body weight loss and weight maintenance in relation to habitual caffeine intake and green tea supplementation. Obes Res. 2005 Jul;13(7):1195-204. doi: 10.1038/oby.2005.142. PMID 16076989
- [Background] Yoshioka M, Doucet E, Drapeau V, Dionne I, Tremblay A. Combined effects of red pepper and caffeine consumption on 24 h energy balance in subjects given free access to foods. Br J Nutr. 2001 Feb;85(2):203-11. doi: 10.1079/bjn2000224. PMID 11242488